CLINICAL TRIAL: NCT01418027
Title: Combined Intensive and Conventional Exercise Intervention of Nonalcoholic Fatty Liver Disease
Brief Title: Combined Intensive and Conventional Exercise on Nonalcoholic Fatty Liver Disease (NAFLD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Xiao-Ying Li, Professor, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CCEMD011
Record Dates: First submitted 2011-08-15; First posted 2011-08-16 (Estimated); Last update posted 2014-09-01 (Estimated); Status verified 2014-08

CONDITIONS: Non-alcoholic Fatty Liver Disease (NAFLD)
Keywords: NAFLD; exercise; hepatic triglycerides
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Intensive exercise (Experimental): The subjects receive an intensive exercise for 6 months and a subsequent conventional exercise for another 6 months.
  Interventions: Other: Intensive exercise
- Lifestyle counseling (No Intervention): Subjects receive a general lifestyle counseling for 12 months
- Regular exercise (Experimental): Subjects receive conventional exercise for 12 months
  Interventions: Other: Conventional exercise

INTERVENTIONS:
Other: Intensive exercise — Subjects conduct an aerobic exercise at 65-80% maximum oxygen consumption for 30 minutes each day, five days a week, totally for 6 months.Subsequently, moderate physical activity(3.0-6.0 MET s) at 150 min/wk for 6 months.
  Arms: Intensive exercise
Other: Conventional exercise — Subjects receive moderate physical activity(3.0-6.0 MET s) at 150 min/wk(30 min per day, five days a week) for 12 months.
  Arms: Regular exercise

SUMMARY:
The prevalence of NAFLD is 50-70% in obese people. A decrease of calorie intake and increase of physical activity are recommended as an effective approach for the prevention and treatment of NAFLD. However, the exercise model for NAFLD intervention is understudied. In the present study we aim to compare the effect of intensive and conventional exercise interventions on NAFLD.

ELIGIBILITY:
1. Subjects with NAFLD determined by MRS ;
2. Age 40-65 years old;
3. Waist circumference> 90cm for men and > 85cm for women.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2011-08; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Change of intrahepatic triglyceride contents | 12 months

SECONDARY OUTCOMES:
Change of body weight | 12 months
Change of waist circumference | 12 months
Change of body fat | 12 months
Change of abdominal fat | 12 montshs
Change of carotid intima-media thickness | 12 months
Change of cardiovascular risk factors (Blood pressure, lipids, glucose) | 12 months
Change of insulin resistance | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoying Li, MD,PhD, Principal Investigator — Shanghai Jiao Tong University School of Medicine
Locations (1):
- The First Hospital Affiliated to Xiamen University, Xiamen, China

REFERENCES:
- [Derived] Zhang HJ, He J, Pan LL, Ma ZM, Han CK, Chen CS, Chen Z, Han HW, Chen S, Sun Q, Zhang JF, Li ZB, Yang SY, Li XJ, Li XY. Effects of Moderate and Vigorous Exercise on Nonalcoholic Fatty Liver Disease: A Randomized Clinical Trial. JAMA Intern Med. 2016 Aug 1;176(8):1074-82. doi: 10.1001/jamainternmed.2016.3202. PMID 27379904